CLINICAL TRIAL: NCT05229523
Title: Validity and Reliability of the Modified Four Square Step Test (mFSST) in Children With Cerebral Palsy
Brief Title: Validity and Reliability of the Modified Four Square Step Test (mFSST)
Acronym: cp
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSUFTR2
Record Dates: First submitted 2022-01-16; First posted 2022-02-08 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy; Diplegic Cerebral Palsy; Hemiplegic Cerebral Palsy; Gait Disorders, Neurologic; Gait, Spastic; Gait Disorders in Children
Keywords: Cerebral Palsy; gait; Modified Four Square Step Test (mFSST); reliability; validity
MeSH Terms: conditions — Cerebral Palsy; Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Children with diparetic and hemiparetic cerebral palsy: 1/Children with diparetic and hemiparetic cerebral palsy aged 7-18 years with the Communication Function Classification System (CFCS) level ≤ 3 and Extended Gross Motor Function Classification System (GMFCS-E&R) level ≤ 2
  Interventions: Other: repeated assessments

INTERVENTIONS:
Other: repeated assessments — validity and reliability of the Modified Four Square Step Test (mFSST) in children with cerebral palsy with the tests of Pediatric Berg Balance Scale (PBSS), Timed Up and Go Test (TUG), Pediatric Functional Reaching Test (PFUT)
  Other Names: validity and reliability of the Modified Four Square Step Test (mFSST) in children with cerebral palsy

SUMMARY:
Cerebral Palsy (CP) is a non-progressive neurodevelopmental disorder that causes activity limitation resulting from movement and posture deficiencies as a result of a lesion in the immature brain. Children with CP usually have difficulties in mobility, transfer and social participation due to many motor and sensory disorders such as muscle weakness, decreased postural control, balance, spasticity.Hypertonus and abnormal motor patterns, lack of trunk control and postural disorders adversely affect the physical development of these children. Children with CP show various posture disorders due to proximal muscle strength losses leading to limitations and deficiencies in postural reactions. This leads to losses in reactive and antisipatory postural adjustments, and limits upper extremity functions such as walking, reaching, and eating. For this reason, children with CP have difficulties in maintaining balance while standing or sitting independently, walking, maintaining postural control in various environments such as walking, hills/uneven floors, performing activities of daily living (ADL) and social participation.

DETAILED DESCRIPTION:
SP; classified as spastic, dyskinetic, ataxic type. The most common type is the spastic type. The ones with the best functional independence level in this group are; hemiparetic and diparetic SP. In addition to the lower extremities, the upper extremities are affected to a small extent in spastic diparetic CP. Increased lower extremity hypertonus in these children causes gait disturbances and balance problems such as fingertip, jumping, scissoring, bent knee gait. In patients with hemiparetic CP, on the other hand, hypertonus, spasticity, inadequacy in trunk control and motor losses are usually observed in one half of the body. In hemiparetic patients, the upper extremity is usually more affected than the lower extremity, and gait pathologies and balance problems are seen in different patterns. Abnormal gait patterns and balance problems are common and common problems in children with CP. As children grow, these disorders in gait become more pronounced as a result of increased hypertonus due to their taller growth. In addition, increased hypertonus and stretch reflex, muscle weakness, coactivation of antagonist muscles, posture disorders, proprioception losses, muscle and joint deformities are other factors that cause gait disorders and balance problems in these children. At this point, the main purpose of CP rehabilitation is to ensure that the child gains maximum functional independence by achieving optimal developmental potential. Therefore, balance and gait restrictions are important problems in children with CP. For these reasons, the evaluation of gait and balance is of great importance in terms of determining the effectiveness of the physiotherapy program, shaping the program, planning and determining the effectiveness of orthopedic and surgical applications, especially in children with CP who have walking potential. In the literature, gait pathologies in children with CP and easy-to-use, valid and reliable observational gait analyzes that can evaluate gait in the clinic are emphasized. These measurements are of great importance in clinical practice. Gait analysis systems including computerized kinetics and kinematics laboratories, electromyography (EMG) and video imaging are the "gold standard" methods used to evaluate the gait of children with CP. However, these evaluation methods are not routinely used in clinics because they are complex, expensive, time-consuming and not easy to apply.On the other hand, performance tests commonly used in the clinic such as the Timed Up and Go Test (TUG), the Timed Up and Down Stairs Test, the 2 Minute Walk Test, and the 6 Minute Walk Test evaluate the functionality of walking. All these tests are tests that evaluate gait prospectively and cannot fully address the child's functional status and balance problems. Therefore, in order to gain and maintain functional independence, the gait problems of the child with CP need to be examined more. In this respect, with a test such as the Modified Four-Square Step Test (mFSST), it provides a different task than normal by assessing the sustainability of postural control, which provides balance parameters by changing direction, and enables the observation of body perception, trunk stability provided by anterior-posterior cocontraction, balance, correction and protective reactions. It is performed using tape instead of canes, according to the Four Square Step test (FSST), which is frequently used in SP and found to be valid and reliable. The mFSST, a modified version of the FSST, could allow more children with CP with balance problems to complete the test while retaining the essential components of obstacle avoidance and the need for individuals to step forward, backward, and to either side. In this test, while passing over an object, the height of the object is reduced. The aim of the study is to examine the validity and reliability of the Modified Four Square Step test (mFSST) in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CP according to SCPE criteria
* Expanded Gross Motor Function Classification System (GMFCS-E&R) Level ≤ 2
* Children aged 7-18 with CP with a Communication Function Classification System (CFCS) ≤ 3
* Children with a Modified Ashworth Scale (MASH) ≤ 3
* Passive range of motion in the ankle, knee and hip joints
* Individuals with spastic hemiparetic-diparetic CP who can follow verbal commands
* Volunteer to participate in the study

Exclusion Criteria:

* Not having had Botox (Botulinum toxin) or surgery in the last 6 months
* Contracture of ankle and knee joint
* Individuals with hemiparetic-diparetic CP who can follow verbal commands

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with spastic diparetic and hemiparetic cerebral palsy
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Modified Four Square Step Test (mFSST) | day 1 (observer1)
  It aims to assess dynamic balance and step objects forward, sideways and backwards. The square drawn on the floor is divided by tape into 4 equal parts. The number 1 is written in the lower right corner, and it is written up to 4 in a clockwise direction. With the start command, individuals are asked to step on the numbers in order. First of all, he is asked to take a step forward (to the number 1 and 2), then to the left (to the number 3), then back to the number (4). He is then asked to take steps from 4 to 1 again. The time is recorded. High time indicates worse dynamic stability.
Modified Four Square Step Test (mFSST) | day 1 (observer2)
  It aims to assess dynamic balance and step objects forward, sideways and backwards. The square drawn on the floor is divided by tape into 4 equal parts. The number 1 is written in the lower right corner, and it is written up to 4 in a clockwise direction. With the start command, individuals are asked to step on the numbers in order. First of all, he is asked to take a step forward (to the number 1 and 2), then to the left (to the number 3), then back to the number (4). He is then asked to take steps from 4 to 1 again. The time is recorded. High time indicates worse dynamic stability.
Modified Four Square Step Test (mFSST) | day 2 (observer2)
  It aims to assess dynamic balance and step objects forward, sideways and backwards. The square drawn on the floor is divided by tape into 4 equal parts. The number 1 is written in the lower right corner, and it is written up to 4 in a clockwise direction. With the start command, individuals are asked to step on the numbers in order. First of all, he is asked to take a step forward (to the number 1 and 2), then to the left (to the number 3), then back to the number (4). He is then asked to take steps from 4 to 1 again. The time is recorded. High time indicates worse dynamic stability.
Modified Four Square Step Test (mFSST) | day 2 (observer1)
  It aims to assess dynamic balance and step objects forward, sideways and backwards. The square drawn on the floor is divided by tape into 4 equal parts. The number 1 is written in the lower right corner, and it is written up to 4 in a clockwise direction. With the start command, individuals are asked to step on the numbers in order. First of all, he is asked to take a step forward (to the number 1 and 2), then to the left (to the number 3), then back to the number (4). He is then asked to take steps from 4 to 1 again. The time is recorded. High time indicates worse dynamic stability.
Pediatric Berg Balance Scale (PBBS) | day 1 (observer1)
  The test has 14 items of increasing difficulty to test functional skills related to activities of daily living, from sitting to standing on one leg. Each item is scored on a five-point ranking scale ranging from 0 to 4 points, with a maximum score level of 56. A higher score indicates better postural balance.
Timed Up and Go Test (TUG) | day 1 (observer1)
  It is a reliable test that measures walking speed, postural control, functional mobility and balance. For the test, the child is seated in a height-adjustable chair. The chair height is adjusted so that the child's feet are in contact with the floor and the knees and hips are flexed to 90 degrees. A distance of 3 meters is marked. When the command is given, the child is asked to get up, walk, return and sit on the chair until the marked area. By starting the time with the start command, the time until sitting is recorded. This test will be repeated 3 times and the average time will be recorded. Increasing time indicates worse balance.
Pediatric Functional Reach test (PFRT) | day 1 (observer1)
  Necessary environmental conditions are provided away from external stimuli. Then, the child is asked to stand sideways on a wall, with the elbows extended in 90 degrees shoulder flexion without touching the wall. The first measurement is made in this position. Then, he is asked to reach forward without taking a step. The last point it can reach is recorded. The distance between these two distances is measured in meters and recorded. The test is repeated when stepping or stopping the contact of the foot with the ground. Increasing the measured distance indicates worse balance.
Four Square Stepping Test (FSST) | day 1 (observer1)
  The child stands in square 2 facing square 1 in a marked area divided into 4 squares. The child has to take turns stepping on each square as fast as possible: it requires the child to step forward, backward, right, and left in a sequence of 2, 3, 4, 1, 4, 3, 2, and 1, respectively. The necessary equipment is a stopwatch and 4 walking sticks 90 cm long. A square with 4 is formed by laying the canes flat on the ground. If the child fails to complete the series, loses balance, or touches the cane during the trial, the trial is repeated. Timing begins with the first foot touching the floor in frame 1 and ends with the last foot touching the floor in frame 4. Test performance is measured in seconds (sec) and shorter completion time means better dynamic stability.

SECONDARY OUTCOMES:
Expanded and revised Gross Motor Function Classification System (GMFCS-E&R) | day 1 (observer1)
  It is a standard classification system used to classify gross motor functions of children with CP. GMFCS classifies levels I to V. Level I indicates the best and V the worst level of motor function.
Modified Ashworth Scale (MAS) | day 1 (observer1)
  It is a method used to determine the severity of spasticity. It is based on the subjective rating of the resistance felt during the examination. Spasticity of the bilateral hip adductors, hip flexors, knee flexors, ankle plantar flexors (gastro-solues) muscles in the lower extremity will be evaluated once at the beginning of the treatment program. The tone felt in these muscles against passive movement is classified as follows; 0: No increase in tone, 1: Slight increase in tone characterized by catching and relaxation or mild resistance at the end of the ROM, 1+: Slight increase in tone characterized by minimal resistance in the remaining ROM (less than half) after capture, 2: Significant tone over most of the ROM increase, but the involved joint can be moved easily, 3: Significant increase in muscle tone, passive movement is difficult, 4: The involved part is rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No